CLINICAL TRIAL: NCT04143204
Title: Early Nutritional Intake and Growth in Very Preterm or Very Low Birth Weight Infants: a Prospective Cohort Study
Brief Title: Nutrition and Growth in Very Preterm Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: NGPI2019
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Premature; Growth
MeSH Terms: conditions — Premature Birth | interventions — Eating; Insulin-Like Growth Factor I; Leptin; Ghrelin; C-Peptide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- very preterm infants cohort: A prospective cohort of very preterm or very low birth weight infants from birth to corrected age 18 months.
  Interventions: Other: Oral nutritional intake

INTERVENTIONS:
Other: Oral nutritional intake — The exposure are oral nutritional intake and all nutritional intake during early life (28 days), and insulin-like growth factor 1, leptin, Ghrelin, and C-peptide in serum at corrected age 40 gestational weeks.
  Other Names: All nutritional intake; Insulin-like growth factor 1; Leptin; Ghrelin; C-peptide

SUMMARY:
This study aims to explore the relation of early nutritional intake, especially oral nutrition intake, with growth and body composition among very preterm or very low birth weight infants.

DETAILED DESCRIPTION:
As the survival of very preterm infants increases, it is important to evaluate their long-term outcomes. Nutritional intake during early life was important to the growth and development in infants, especially in preterm infants. Studies found that early nutrition exposure in preterm infants can effect scored of Griffith Mental Development Scales and body fat percentage at later life. Insulin-like growth factor-1, leptin, Ghrelin, C-Peptide are associated with fat mass in children. And accumulation of fat and insulin resistance (IR) in the early postnatal period are related to metabolism diseases in adulthood. However, previous studies on nutrition and growth or the body composition of preterm infants were mostly completed in developed countries, and no relevant data were available in China. Therefore, this study aims to establish a prospective cohort of very preterm infants to observe the effects of nutritional exposure in early life on growth and body composition in later life.

ELIGIBILITY:
Inclusion Criteria:

* infants born with a gestational age >=28 weeks and <32 weeks and/or a birth weight >=1000g and <1500g;
* infants admitted to neonatal intensive care unit (NICU) of Children's hospital of Fudan University within 24h after birth.

Exclusion Criteria:

* major congenital anomalies or heredity metabolic diseases;
* severe disease or abdominal surgery during hospitalization;
* death during hospitalization or discharge without medical advice;
* small for gestational age.

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very preterm or very low birth weight infants in NICU
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Z-scores of weight | at corrected age 40 gestational weeks
  Computed according to the Fenton preterm growth standards (2013)

SECONDARY OUTCOMES:
Z-scores of length/height | at corrected age 40 gestational weeks
  Computed according to the Fenton preterm growth standards (2013)
Z-scores of head circumference | at corrected age 40 gestational weeks
  Computed according to the Fenton preterm growth standards (2013)
Z-scores of weight | at corrected age 6 months and 18 months
  Computed according to the WHO standards (2006)
Z-scores of length/height | at corrected age 6 months and 18 months
  Computed according to the WHO standards (2006)
Z-scores of head circumference | at corrected age 6 months and 18 months
  Computed according to the WHO standards (2006)
Percentage of infants who achieve catch-up growth | at corrected age 6 months and 18 months
  Catch-up growth is defined as weight, length/height or head circumference equal to or above the 25th percentile for corrected age, according to the WHO standards (2006).
Body fat free mass | at corrected age 40 gestational weeks and 6 months
  assessed by air displacement plethysmography (ADP)
Body fat mass | at corrected age 40 gestational weeks and 6 months
  assessed by air displacement plethysmography (ADP)
Body fat proportion | at corrected age 40 gestational weeks and 6 months
  assessed by air displacement plethysmography (ADP)
Cognitive development outcome | at corrected age 18 months
  It is examined by six areas of development measured by Griffith Mental Development Scales (GMDS) including locomotor, personal-social, hearing and language, eye and hand co-ordination, performance and practical reasoning. Developmental impairment is defined as a developmental quotient lying one standard deviation below the mean (<85) and includes mild impairments (70-84) and moderate/severe impairment (<70).
Intestinal flora change | from birth to corrected age 18 months
  The change of composition of intestinal flora in preterm infants. The composition of intestinal flora was test by 16s rRNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Yan, MD, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No